CLINICAL TRIAL: NCT07135986
Title: A Phase 3, Modified Double-blind, Multi-center Study of the Immunogenicity and Safety of an Investigational Quadrivalent Meningococcal Conjugate Vaccine Administered in Healthy Children and Adolescents (2 to 17 Years of Age) in China
Brief Title: Immunogenicity and Safety Study of an Investigational Quadrivalent Meningococcal Conjugate Vaccine Administered in Healthy Children and Adolescents in China
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MEQ00076; U1111-1256-8979 (Registry Identifier: ICTRP)
Record Dates: First submitted 2025-08-14; First posted 2025-08-22 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Meningococcal Infection; Healthy Volunteers
MeSH Terms: conditions — Meningococcal Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Investigators and study staff as well as Sponsor study staff who conduct the safety assessment and the participant/parent/LAR will not know which study intervention is administered. Only the study staff who prepare and administer the study intervention and are not involved with the safety evaluation will know which study intervention is administered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Group 1 MenACYW1-dose schedule (Experimental): 1 dose of MenACYW conjugate vaccine to participants aged 7 through 17 years of age
  Interventions: Biological: MenACYW conjugate vaccine
- Group 2 MenACYW135 Ps 1-dose schedule (Active Comparator): 1 dose of MenACYW135 polysaccharide vaccine to participants aged 7 through 17 years of age
  Interventions: Biological: MenACYW135 polysaccharide vaccine
- Group 3 MenACYW1-dose schedule (Experimental): 1 dose of MenACYW conjugate vaccine to participants aged 2 through 6 years of age
  Interventions: Biological: MenACYW conjugate vaccine
- Group 4 Royal MenAC1-dose schedule (Active Comparator): 1 dose of Royal's MenAC conjugate vaccine to participants aged 2 through 6 years of age
  Interventions: Biological: MenAC conjugate vaccine

INTERVENTIONS:
Biological: MenACYW conjugate vaccine — Pharmaceutical form:Liquid solution-Route of administration:Intramuscular (IM) injection
  Other Names: MenQuadfi
  Arms: Group 1 MenACYW1-dose schedule; Group 3 MenACYW1-dose schedule
Biological: MenACYW135 polysaccharide vaccine — Pharmaceutical form: Lyophilized powder-Route of administration:IM injection
  Arms: Group 2 MenACYW135 Ps 1-dose schedule
Biological: MenAC conjugate vaccine — Pharmaceutical form:Lyophilized powder-Route of administration:IM injection
  Arms: Group 4 Royal MenAC1-dose schedule

SUMMARY:
This is a Phase 3, modified double-blind, randomized, parallel-group, active-controlled, multicenter study with 2 arms and 4 groups to evaluate the immunogenicity and safety of MenACYW conjugate vaccine in children and adolescents versus control meningococcal vaccines licensed in China.

Study details include:

* The study duration will be approximately 180 days.
* The vaccination visit will be Visit 1.
* The visit frequency will be 2 on-site visits with a 30-day interval. A safety visit/telephone call is planned on the ninth day after the vaccination for all groups; a safety follow-up telephone call is planned for all groups 180 days post the last vaccination.

DETAILED DESCRIPTION:
The duration of each participant's participation will be approximately 180 days.

ELIGIBILITY:
Inclusion Criteria:

* For Cohort I: Aged 7 to 17 years on the day of inclusion ("7 to 17 years" means from the day of the 7th birthday to the day before the 18th birthday.). For Cohort II: Aged 2 to 6 years on the day of inclusion (2 to 6 years" means from the day of the 2nd birthday to the day before the 7th birthday.)
* Participants who are healthy as determined by medical evaluation including medical history and physical examination.
* A female participant is eligible to participate if she is not pregnant or breastfeeding

Exclusion Criteria: Participants are excluded from the study if any of the following criteria apply:

* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy; or long-term systemic corticosteroid therapy
* History of meningococcal infection
* History of any neurologic disorders
* History of Guillain-Barré syndrome
* History of an Arthus-type hypersensitivity reaction after a previous dose of tetanus toxoid-containing vaccine
* At high risk for meningococcal infection during the trial
* Known systemic hypersensitivity to any of the vaccine components
* Self-reported thrombocytopenia, contraindicating intramuscular vaccination.
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular vaccination.
* Chronic illness that, in the opinion of the Investigator, is at a stage where it might interfere with trial conduct or completion.
* Moderate or severe acute illness/infection
* Alcohol, prescription drug, or substance abuse that, in the opinion of the Investigator, might interfere with the study conduct or completion.
* Receipt of any vaccine in the 4 weeks preceding the trial vaccination or planned receipt of any vaccine in the 4 weeks following trial vaccination.
* The time since last vaccination of meningococcal vaccine was 2 years or less.
* Receipt of immune globulins, blood or blood-derived products in the past 3 months.
* Receipt of oral or injectable antibiotic therapy within 72 hours prior to the first blood draw.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1602 (Estimated)
Dates: Start 2025-09-26 (Actual); Primary Completion 2026-06-05 (Estimated); Study Completion 2026-11-02 (Estimated)

PRIMARY OUTCOMES:
Participants 7 through 17 years of age (Cohort I): Vaccine seroresponse to meningococcal serogroups A, C, Y, and W | Day 01 (pre-vaccination) and Day 31 (post- vaccination)
  30 days postvaccination rSBA titer ≥1:8 for participants with prevaccination rSBA titer <1:8, or At least 4-fold increase in rSBA titer from pre- to 30 days postvaccination for participants with pre vaccination rSBA titer ≥1:8
Participants 7 through 17 years of age (Cohort I): Geometric mean titers (GMTs) of antibodies against meningococcal serogroups A, C, Y, and W | Day 31 (post- vaccination)
  Antibodies titers are expressed as geometric mean titers
Participants 7 through 17 years of age (Cohort I): Vaccine seroresponse to meningococcal serogroups W and Y will be assessed in participants receiving MenACYW conjugate vaccine | Day 01 (pre-vaccination) and Day 31 (post- vaccination)
  30 days postvaccination rSBA titer ≥1:8 for participants with prevaccination rSBA titer <1:8, or At least 4-fold increase in rSBA titer from pre- to 30 days post-vaccination for participants with pre vaccination rSBA titer ≥1:8
Participants 2 through 6 years of age (Cohort II): Vaccine seroresponse to meningococcal serogroups A and C | Day 01 (pre-vaccination) and Day 31 (post- vaccination)
  30 days postvaccination rSBA titer ≥1:8 for participants with prevaccination rSBA titer <1:8, or At least 4-fold increase in rSBA titer from pre- to 30 days postvaccination for participants with pre vaccination rSBA titer ≥1:8
Participants 2 through 6 years of age (Cohort II): Geometric mean titers (GMTs) of antibodies against meningococcal serogroups A and C | Day 01 (pre-vaccination) and Day 31 (post- vaccination)
  Antibody titers are expressed as geometric mean titers
Participants 2 through 6 years of age (Cohort II): Vaccine seroresponse to meningococcal serogroups W and Y in participants receiving MenACYW conjugate vaccine | Day 01 (pre-vaccination) and Day 31 (post- vaccination)
  30 days post-vaccination rSBA titer ≥1:8 for participants with pre-vaccination rSBA titer <1:8, or At least 4-fold increase in rSBA titer from pre- to 30◦days post-vaccination for participants with pre vaccination rSBA titer ≥1:8

SECONDARY OUTCOMES:
Number of participants with immediate adverse events (AEs) | Within 30 minutes post-vaccination
  Unsolicited systemic AEs that occur within 30 minutes after vaccination
Presence of solicited injection site reactions | Within 7 days post-vaccination
  Solicited injection site reactions include injection site pain, erythema and swelling
Presence of solicited systemic reactions | Within 7 days post-vaccination
  Solicited systemic reactions include fever, headache, malaise and myalgia
Presence of unsolicited AEs | Within 30 days post-vaccination
Presence of SAEs | Up to Day 181 post-vaccination
  SAEs, including adverse events of special interest (AESIs), reported throughout the study
Participants 7 through 17 years of age (Cohort I): Antibody titers against meningococcal serogroups A, C, Y, and W in Groups 1 and 2 | Day 01 (pre-vaccination) and Day 31 (post- vaccination)
  Antibody titers measured by rSBA titer ≥1:8, ≥1:128
Participants 2 through 6 years of age (Cohort II): Antibody titers against meningococcal serogroups A, C, Y, and W in Group 3 and against meningococcal serogroups A and C in Group 4 | Day 01 (pre-vaccination) and Day 31 (post- vaccination)
  Antibody titers measured by rSBA titer ≥1:8, ≥1:128
Participants 2 through 6 years of age (Cohort II): Antibody titers in terms of GMTs against meningococcal serogroups Y and W in Group 3 | Day 01 (pre-vaccination) and Day 31 (post- vaccination)
  Antibodies titers are expressed as geometric mean titers

CONTACTS AND LOCATIONS:
Locations (1):
- Investigational Site Number : 1561000, Nanning, Guangxi, China

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: MEQ00076 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=26816&tenant=MT_SNY_9011